CLINICAL TRIAL: NCT02916147
Title: Comparison of Volatile and IV Anesthesia on the Change of Alarmins in Lung Cancer Patients Receiving Pulmonary Lobectomy
Brief Title: Effect of Different Anesthetics on the Change of Alarmins in Lung Cancer Patients Receiving Pulmonary Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: E2016066
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- volatile anesthesia (Experimental): Use 2-3% sevoflurane to maintain the anesthesia during OLV surgery with bispectral index (BIS) 40-60.
  Interventions: Drug: Sevoflurane
- intravenous anesthesia (Active Comparator): Anesthesia was maintained by a continuous infusion of propofol （4-6mg/kg/h）with BIS 40-60.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane
  Arms: volatile anesthesia
Drug: Propofol
  Arms: intravenous anesthesia

SUMMARY:
This study aim to observe and compare the change of alarmins such as high mobility group nucleosome-binding protein-1 (HMGN1), high mobility group proteins b1 (HMGb1), Interleukin (IL)-33 and their soluble receptors including soluble toll like receptor 4 (sTLR4) and soluble ST2 (sST2) during pulmonary lobectomy for cancer patients receiving volatile anesthesia or intravenous anesthesia under one-lung ventilation (OLV). By which, this study will preliminarily evaluate the correlation of alarmins and prognosis as well as the effect of inhalational and intravenous anesthesia on the prognosis of surgical patients.

DETAILED DESCRIPTION:
During pulmonary lobectomy, as a result of OLV and surgical operation, patients can suffer from alveolar and systemic inflammatory response. Alarmin is endogenous peptide released by white blood cells and epithelial cells when the body undergo danger signal stimulation which can enhance immune response and has a double effect on tumor. Some alarmins and their soluble receptors such as HMGN1, HMGb1, IL-33 and their soluble receptors including sTLR4 and sST2 can be used as biomarkers for tumor progression. Previous studies have shown that sevoflurane anesthesia can reduce the level of inflammatory cytokines in bronchoalveolar lavage fluid. Meanwhile, the latest retrospective study indicated that the mortality of cancer patients receiving volatile anesthesia was significantly higher than that of intravenous anesthesia. At this stage, no study aimed to investigate the change of alarmins in broncho-alveoli and serum during OLV lung surgery and the possible effect of different anesthetics on them. Therefore, the investigators plan to enroll 40 patients with lung cancer receiving pulmonary lobectomy. Patients are randomly divided into sevoflurane volatile anesthesia group and propofol intravenous anesthesia group (n=20). Perioperative serum and bronchoalveolar lavage from ventilated lung are obtained, using ELISA method, to assay and compare the changes of alarmins such as HMGN1, HMGb1, IL-33 and their soluble receptors including sTLR4 and sST2 between two groups. All the patients will be followed up for 12 months. The correlation of alarmins and prognosis as well as the effect of volatile and intravenous anesthesia on the prognosis of patients will be preliminarily evaluated.

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesiology (ASA) status I-II
* pathological diagnosis of lung cancer before surgery
* receive pulmonary lobectomy
* with normal lung function
* without heart failure (NYHA>2), obstructive or restrictive lung disease
* no history of other malignancy tumor
* body mass index (Body mass, index, BMI) < 35kg/m2
* no severe coagulopathy
* no severe systemic or pulmonary infection
* did not participate in other clinical trials

Exclusion Criteria:

* persistent smoking history
* immunosuppressive drug use 6 weeks before operation
* receive total pneumonectomy
* failure to complete treatment or follow-up
* severe adverse drug reactions
* severe postoperative complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change of level of HMGN1 | 10 min before OLV, 10 min after OLV, 1 day and 2 day after surgery
Change of level of HMGb1 | 10 min before OLV, 10 min after OLV, 1 day and 2 day after surgery
Change of level of sTLR4 | 10 min before OLV, 10 min after OLV, 1 day and 2 day after surgery
Change of level of IL-33 | 10 min before OLV, 10 min after OLV, 1 day and 2 day after surgery
Change of level of sST2 | 10 min before OLV, 10 min after OLV, 1 day and 2 day after surgery

SECONDARY OUTCOMES:
Disease-free survival | 12 months
  disease-free survival means the amount of time that patient lives without known recurrence after surgery to the end of observation or recurrence.
Overall survival | 12 months
  Overall survival means the amount of time that patient lives to the end of observation or death.

CONTACTS AND LOCATIONS:
Overall Officials: Kaiyuan Wang, PhD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital